CLINICAL TRIAL: NCT02942329
Title: Exploratory Clinical Study of the Combination of Apatinib and SHR-1210 in Treating Advanced Hepatocellular Carcinoma or Gastric Cancer
Brief Title: Exploratory Clinical Study of Apatinib and SHR-1210 in Treating Advanced Hepatocellular Carcinoma or Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APA-01
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer; Hepatocellular Carcinoma
Keywords: humanized anti-PD-1 monoclonal antibody; apatinib; Gastric Neoplasms; Gastric Cancer; Cancer of Stomach; Hepatocellular Carcinoma; Liver Cancer, Adult; Liver Cell Carcinoma
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- apatinib and SHR-1210 (Experimental): Every patients will received apatinib orally every day and SHR-1210 200mg (3mg/kg for underweight patients) iv every 2 weeks until disease progression or intolerance of side effects.
  Interventions: Drug: apatinib; Drug: SHR-1210

INTERVENTIONS:
Drug: apatinib — Apatinib was administered 250mg or 375mg orally daily. For gastric cancer patients, the dose would be 250mg or 375mg daily. For hepatocellular carcinoma patients, the dose would be 250mg daily.
Drug: SHR-1210 — SHR-1210 was administered 200mg (3mg/kg for underweight patients) iv every 2 weeks.

SUMMARY:
The purpose of this study is to observe and preliminary explore the efficacy and safety of combination of Apatinib and SHR-1210 regimen in treating advanced hepatocellular carcinoma or gastric cancer.

Apatinib is a small-molecule vascular endothelial growth factors receptor (VEGFR) tyrosine kinase inhibitor, similar to vatalanib (PTK787), but with a binding affinity 10 times that of vatalanib or sorafenib.

SHR-1210 is a humanized anti-PD-1 monoclonal antibody.

DETAILED DESCRIPTION:
Patients will received apatinib orally every day and SHR-1210 200mg (3mg/kg for underweight patients) iv every 2 weeks. The efficacy and safety will be observed.

The dose escalation phase has completed for apatinib from 125mg, 250mg to 500mg. The dose of 250mg showed best tolerance and efficacy especially in hepatocellular carcinoma. Thus, for hepatocellular carcinoma patients, apatinib 250mg orally every day was chosed for the dose extension phase. In gastric cancer, the dose of 250mg also showed good tolerance but mild efficacy. Thus, for gastric cancer patients, the dose of 375mg daily for apatinib would be explored and then the investigators will decide the best dosage for these patients.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria

1. Aged 18-70 years old, both genders.
2. To be confirmed to meet the clinical diagnosis standard, histologically or cytologically confirmed with hepatocellular carcinoma or gastric cancer. Patients must be diagnosed with advanced disease(not eligible for surgical and/or locoregional therapies, or metastatic disease), disease progressed or refractory to standard therapies(had been intolerant to standard therapies, or had refused standard therapy), or lack of other effective treatment methods.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
4. Life expectancy of at least 3 months.
5. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
6. For patients with advanced hepatocellular carcinoma, liver function status Child-Pugh Class A or B (score<=7).
7. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment)as determined by: Hemoglobin ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L (for patients with advanced hepatocellular carcinoma), Platelet count ≥ 100×109/L (for patients with advanced gastric cancer); serum albumin ≥2.8 g/dL; serum total bilirubin (TBIL)≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal(ULN), for subjects with liver metastases, ALT and AST≤5×ULN; Calculated creatinine clearance (CrCl) > 50 mL/min (Cockcroft-Gault formula will be used to calculate CrCl).
8. Females of childbearing potential (FOCBP), who are not surgically sterile or postmenopausal, must conduct pregnancy test (serum or urine) within 7 days before enrollment, and must not be pregnant or breast-feeding women. If the result is negative, she must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs. And non-sterilized males who are sexually active must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs.
9. Patients join the study voluntarily, sign a consent form, have good compliance, and comply with follow-up.

Exclusion Criteria:

1. Patients must not have had prior treatment with SHR-1210 or any other PD-L1 or PD-1 antagonists, and must not have had be enrolled in the phase III Study of Apatinib After Systemic Therapy in Patients With Hepatocellular Carcinoma.
2. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed.
4. Known history of hypersensitivity to any components of the SHR-1210 formulation, or other antibody formulation.
5. Active central nervous system (CNS) metastases with clinical symptoms (including cerebral edema, steroid requirement, or progressive disease). Subjects with brain or meningeal metastases that were previously treated must be clinically stable (magnetic resonance imaging [MRI] at least 4 weeks apart do not show evidence of new or enlarging metastases) and have discontinued immunosuppressive doses of systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration.
6. Patients with other malignant tumor (except cured skin basal cell carcinoma and cervical carcinoma).
7. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention, left ventricular ejection fraction(LVEF) < 50%.
8. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
9. Coagulation abnormalities (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
10. Prior systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks (Or 5 half-life of the drug, calculate the longer ) before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 (with the exception of any stable chronic toxicities not expected to resolve).
11. Patients with clinical symptoms of ascites or pleural effusion, need therapeutic puncture and drainage.
12. Previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency, such as: esophageal varices, local active ulcerative lesions, gastric ulcer and duodenal ulcer, the ulcerous colitis, gastrointestinal diseases such as portal hypertension or resection of tumor with bleeding risk, etc.
13. Patients with or previous with serious hemorrhage (bleeding > 30 ml within 3 months), haemoptysis (> 5 ml within 4 weeks) of thromboembolic events within 12 months (including stroke events and/or transient ischemic attack).
14. Active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled).
15. Previous experience abdomen fistula, gastrointestinal perforation, or abdominal abscess within 4weeks.
16. Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, pulmonary function damaged seriously etc.
17. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or active hepatitis (transaminase does not meet the inclusion, hepatitis B virus (HBV) DNA ≥10⁴ /ml or hepatitis C virus (HCV) RNA≥103 /ml or higher); Chronic hepatitis B virus carriers who HBV DNA<2000 IU/ml(<104/ml), must receive anti-viral treatment throughout the study.
18. Participated in other clinical trials, or finish other clinical trials within 4 weeks.
19. Patients who may receive other anti-tumor systemic chemotherapy during the study.
20. Patients who has bone metastasis, have received Palliative radiotherapy (radiotherapy area > 5% marrow area).
21. Patients who may receive vaccination during the study, or previous had vaccination within 4 weeks.
22. Mental disorders history, or psychotropic drug abuse history.
23. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | Up to approximately 12 months
  6 months and 12 months

SECONDARY OUTCOMES:
Tumor response rate | Up to approximately 12 months
Disease control rate | Up to approximately 12 months
Duration of response | Up to approximately 12 months
Safety as measured by the rate of AEs, deaths and laboratory abnormalities (e.g. Grade 3 or higher per CTCAE v4 ) | From the first assignment of informed consent form up to 90 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Ming Xu, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Locations (1):
- The Affiliated Hospital of the Chinese Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638